CLINICAL TRIAL: NCT03266952
Title: Stroke Incidence and Risk Factors in a Tri-ethnic Region
Acronym: NOMAS
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Columbia University (Other)
Responsible Party: Principal Investigator, Ralph L Sacco, MD MS, Principal Investigator, University of Miami
Other Study IDs: 20070212; R37NS029993 (NIH)
Record Dates: First submitted 2017-08-26; First posted 2017-08-30 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Diabetes; Diet; Epidemiology; Stroke; Myocardial Infarction
Keywords: stroke; race; diet; diabetes; ethnicity; myocardial infarction
MeSH Terms: conditions — Diabetes Mellitus; Stroke; Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Enrollment of a population-based, prospective cohort of 3298 stroke-free adults was completed in 2001 and annual follow-up has continued since then. This collaborative study is the first prospective cohort study among whites, blacks and Caribbean Hispanics living in the same community. This grant supports continued follow-up and outcome detection and expansion of data collection in this cohort. The aims are to evaluate the relationship between vascular outcomes (stroke, myocardial infarction (MI), and vascular death) and insulin resistance, carotid intima-media thickness, carotid distensibility, and quantitative magnetic resonance imaging (MRI) measures of vascular subclinical brain disease and to determine if MRI subclinical disease accounts for race/ethnic differences in cognitive impairment. To accomplish these aims further data collection using the population-based, prospective cohort study is proposed. Stored baseline serum will be used to measure fasting insulin levels to evaluate insulin resistance. High-resolution carotid imaging data will be collected at subsequent visits to expand the measurements of subclinical carotid disease to 1300 subjects. MRIs and a neuropsychological battery emphasizing frontal executive domains will be done on 1300 subjects and quantitative analyses performed to measure white matter hyperintensities, silent infarcts, and silent cerebral microbleeds.

Starting in 2005, subjects enrolled in the MRI substudy began to have echocardiograms and 24hour ambulatory blood pressure monitoring. Subjects will be followed by annual telephone interviews to ascertain stroke, MI, death, and changes in cognitive state. In-person assessment will be done for all subjects who screen positive. Community stroke surveillance will be maintained to insure stroke detection among the cohort. Specific diagnostic committees classify stroke, MI and vascular death.

DETAILED DESCRIPTION:
Stroke remains a major public health problem with a disproportionate impact on blacks and Hispanics.

Studies in Northern Manhattan have demonstrated that blacks and Hispanics have a greater stroke incidence and more frequently have small vessel and intracranial atherosclerotic stroke than whites.

The reasons for these race/ethnic disparities are not entirely clear. Enrollment of a population-based, prospective cohort of 3298 stroke-free adults was completed in 2001 and annual followup has continued since then. This collaborative study is the first prospective cohort study among whites, blacks and Caribbean Hispanics living in the same community. This grant supports continued followup and outcome detection and expansion of data collection in this cohort. The aims are to evaluate the relationship between vascular outcomes (stroke, MI, and vascular death) and insulin resistance, carotid intima-media thickness, carotid distensibility, and quantitative MRI measures of vascular subclinical brain disease and to determine if MRI subclinical disease accounts for race/ethnic differences in cognitive impairment. To accomplish these aims further data collection using the population-based, prospective cohort study is proposed. Stored baseline serum will be used to measure fasting insulin levels to evaluate insulin resistance. High resolution carotid imaging data will be collected at subsequent visits to expand the measurements of subclinical carotid disease to 1300 subjects. MRIs and a neuropsychological battery emphasizing frontal executive domains will be done on 1300 subjects and quantitative analyses performed to measure white matter hyperintensities, silent infarcts, and silent cerebral microbleeds.

Starting in 2005, subjects enrolled in the MRI substudy began to have echocardiograms and 24hour ambulatory blood pressure monitoring. Subjects will be followed by annual telephone interviews to ascertain stroke, MI, death, and changes in cognitive state. In-person assessment will be done for all subjects who screen positive. Community stroke surveillance will be maintained to insure stroke detection among the cohort. Specific diagnostic committees classify stroke, MI and vascular death. The strengths of this cohort study are the wealth of baseline data already assembled, the triethnic composition residing in the same community, the outstanding followup record, the evaluation of putative risk factors, and the innovative assessment of MRI subclinical disease and carotid subclinical disease. The study primary hypotheses are:1. To determine the independent association of insulin resistance among nondiabetics and the incidence of stroke, as well as stroke, MI or vascular death, after adjusting for known modifiable risk factors such as hypertension, lipids, cigarettes, and alcohol. 2.

To evaluate the independent association of subclinical carotid disease (carotid intima-media thickness and carotid distensibility) and the incidence of stroke, MI or vascular death after adjusting for conventional modifiable vascular risk factors, as well as novel vascular risk factors such as homocysteine, high density lipoprotein (HDL) subpopulations, and insulin resistance.3. To compare the prevalence of subclinical vascular brain disease as measured by quantitative MRI, including white matter hyperintensities, silent infarcts, and silent cerebral microbleeds, in each race/ethnic subgroup and determine the association between subclinical brain disease and modifiable vascular risk factors measured up to 10 years prior to MRI. Vascular risk factors will include baseline and repeated measures of conventional modifiable conditions such as hypertension, diabetes, lipid levels, cigarette smoking, physical activity, alcohol use, as well as less-well documented factors such as homocysteine, HDL subpopulations, and insulin resistance. 4. To determine the relationship between subclinical vascular brain diseases and cognitive impairment, particularly diminished performance in frontal executive tests, and whether these MRI findings help explain cognitive performance differences among whites, blacks and Hispanics after adjusting for age and education.5. To explore whether subclinical vascular brain diseases are important predictors of stroke, MI or vascular death. Beginning in Summer 2005, some new aims were added as follows: 1) to determine whether aortic arch abnormalities and/or cardiac abnormalities, and/or 24hour blood pressure levels and changes, are independently associated with silent brain infarcts in the elderly; 2) to determine the risk of symptomatic stroke, myocardial infarction and vascular death associated with aortic/cardiac/24hour blood pressure abnormalities. As of 2010 the investigators will be collaborating with other institutions under the NINDS Ischemic Stroke Genetics (ISG) study. The aims of the NINDS Ischemic Stroke Genetics Study (NINDS ISG Study; NIH Grant 1 U01 NS06920801) are to:1) Assemble ischemic stroke phenotypic data and high quality DNA data from 10 stroke studies. (Participating studies in the NINDS ISG Study: Ischemic Stroke Genetics Study; Siblings with Ischemic Stroke Study; Greater Cincinnati/Northern Kentucky Stroke Study; Genes Affecting Stroke Risk and Outcome Study/Bugher Network Study; Northern Manhattan Study; Baltimore/Washington Young Stroke Study; Heart and Vascular Health Stroke Study; Nurses Health Study; Reasons for Geographic and Racial Differences in Stroke; Women's Health Initiative). This collaboration has access to 7,033 cases of ischemic stroke and 23,411 study-specific controls. 2) Test for associations with ischemic stroke and its subtypes in the NINDS ISG Study. 3) Replicate and extend associations detected in Aim 1.2 above by taking advantage of other genomewide association studies conducted by other members of the Ischemic Stroke Genetics studies.

ELIGIBILITY:
Inclusion Criteria:

* Northern Manhattan Study participants were selected using random-digit dialing with the following eligibility criteria: never diagnosed with stroke; greater than 40 years old; resided in Northern Manhattan for at least 3 months, in a household with a telephone.

Exclusion Criteria:

* For this analysis we excluded participants with diabetes mellitus at baseline, defined by the participant's self-reported diabetes, use of insulin or oral anti-diabetic medication, or fasting glucose at least 126 mg/dl. We also excluded participants missing data for soda consumption, and those with improbable total daily kilocalories based on food frequency responses.

Min Age: 40 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NOMAS is a prospective population-based cohort study, recruited 1993-2001, with the original goal of identifying the incidence of and risk factors for stroke in a multi-ethnic urban adult population. Northern Manhattan is a well-defined region of New York City with a race/ethnic distribution of 63% Hispanics, 20% Non-Hispanic black, and 15% non-Hispanic white residents
Sampling Method: Probability Sample
Enrollment: 3497 (Actual)
Dates: Start 1993-01 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Incidence of Stroke | 24 years
  Stroke is defined as first symptomatic stroke of any type, based on World Health Organization (WHO) criteria as "rapidly developing clinical signs of focal (at times global) disturbance of cerebral function, lasting more than 24 hours or leading to death with no apparent cause other than that of vascular origin"

SECONDARY OUTCOMES:
Incidence of myocardial infarction | 24 years
  Myocardial Infarction is defined using the clinical, ECG and cardiac enzyme criteria adapted from the Cardiac Arrhythmia Suppression Trial and the Lipid Research Clinics Coronary Primary Prevention Trial and requires at least 2 of the 3 following criteria: (a) ischemic cardiac pain; (b) cardiac enzyme abnormalities; and (c) ECG abnormalities.
Incidence of vascular death | 24 years
  Death is classified as either being of vascular nature if due to stroke, myocardial infarction, heart failure, pulmonary embolus, or cardiac arrhythmia to the extent that this can be determined from available records and sources
Scoring cognitive impairment | Mean of 6 years after baseline
  A neuropsychological battery was administered and participants were scored on 4 cognitive domains: semantic memory, episodic memory, executive function, processing speed

OTHER OUTCOMES:
Incidence of diabetes | 24 years
  Self-reported incidence of diabetes

CONTACTS AND LOCATIONS:
Overall Officials: Ralph L Sacco, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No